CLINICAL TRIAL: NCT00477100
Title: Inflammatory Breast Cancer (IBC) Registry
Brief Title: Biospecimen and Medical Data Collection and Tumor Biopsy in Creating Research Tissue Registry in Patients With Inflammatory or Invasive Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Texas Appropriation for Rare and Aggressive diseases (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2006-1072; NCI-2018-01784 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006-1072 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Breast Carcinoma; Invasive Breast Carcinoma; Second Primary Malignant Neoplasm
MeSH Terms: conditions — Inflammatory Breast Neoplasms; Neoplasms, Second Primary | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen and medical data collection): Patients complete questionnaires and participate in interview over 30 minutes. Patients also undergo collection of medical data and blood, tissue, and stool samples.
  Interventions: Procedure: Biospecimen Collection; Other: Interview; Other: Medical Chart Review; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, tissue, and stool
Other: Interview — Participate in interview
Other: Medical Chart Review — Undergo collection of medical data
  Other Names: Chart Review
Other: Questionnaire Administration — Ancillary Studies

SUMMARY:
This trial studies the biospecimen and medical data collection in creating a research tissue registry in patients with inflammatory or invasive breast cancer. Collecting medical data and storing samples of blood, tissue, and stool from patients with inflammatory breast cancer to study in the laboratory may help doctors find better ways to treat and study inflammatory breast cancer in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively collect tissue (including primary inflammatory breast cancer [IBC], ipsilateral nodal metastasis and/or distant metastasis [if applicable] obtained prior to primary systemic therapy and mastectomy/axillary dissection), serum, plasma, whole blood, clinical, and imaging data from patients with recently diagnosed inflammatory breast cancer (IBC), or highly suspicious for IBC, who have not received systemic therapy.

II. To collect paraffin tissue blocks or unstained slides (including primary, ipsilateral nodal metastasis and/or distant metastasis [if applicable] obtained prior to primary systemic therapy), mastectomy/axillary dissection tissue, serum, plasma, whole blood, clinical, and imaging data (if available) from patients with previously diagnosed inflammatory breast cancer (IBC), who have been treated or partially treated, but have not had mastectomy and are seeking further treatment in the IBC clinic at M. D. Anderson or participating cancer network sites.

III. To collect oral swab, skin and stool bacterial culture swab for microbiome analysis to compare patients with specific breast cancer subtype to report changes in flora during the course of treatment and correlated to toxicity.

OUTLINE:

Patients complete questionnaires and participate in interview over 30 minutes. Patients also undergo collection of medical data and blood, tissue, and stool samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of primary inflammatory breast cancer (IBC), second primary IBC, or highly suspicious for IBC (MD Anderson patients only).
* Histological diagnosis of invasive breast cancer, or highly suspicious for IBC (MD Anderson patients only) but pending breast cancer diagnosis.
* Be either newly diagnosed, or highly suspicious for IBC (MD Anderson patients only) [Cohort I] or have paraffin blocks or up to 20 unstained slides of each representative block(s) from the time of initial diagnosis of IBC(i.e. core biopsy and punch biopsy) and/or from mastectomy (Cohort II-MD Anderson patients only)
* Age > 18 years
* Able to provide informed consent

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with inflammatory or invasive breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2007-04-17 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Data, serum, tissue, peripheral blood mononuclear cells, and plasma sample collection | Up to 2 years
  No statistical considerations are provided. For each clinical question that will use the data collected in this registry, a separate protocol will be submitted to the Institutional Review Board (IRB) that will include a sample size justification and an analysis plan.

CONTACTS AND LOCATIONS:
Overall Officials: VIcente Valero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (10):
- United States (10):
  - Banner - MD Anderson Cancer Center, Gilbert, Arizona
  - Scripps - MD Anderson Cancer Center, La Jolla, California
  - Banner - MD Anderson Cancer Center - Northern Colorado, Greeley, Colorado
  - Baptist - MD Anderson Cancer Center, Jacksonville, Florida
  - Covenant Medical Center, Saginaw, Michigan
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - MD Anderson League City, Nassau Bay, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - MD Anderson in The Woodlands, The Woodlands, Texas

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org